CLINICAL TRIAL: NCT02072473
Title: Safety and Efficacy Aspects of a Standardized Stepwise Anatomical Approach for Atrio-Ventricular Nodal Re-entrant Tachycardia Ablation
Brief Title: Safety and Efficacy Aspects of a Standardized Stepwise Anatomical Approach for AVNRT Ablation
Status: Withdrawn | Type: Observational
Why Stopped: No enrollment
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: SHEBA-0716-13-RB-CTIL
Record Dates: First submitted 2014-02-10; First posted 2014-02-26 (Estimated); Last update posted 2016-10-19 (Estimated); Status verified 2016-10

CONDITIONS: Re-entrant Atrioventricular Node Tachycardia
Keywords: Re-entrant Atrioventricular Node Tachycardia; Unsuccessful right-sided slow pathway ablation; Coronary sinus / left-sided slow pathway ablation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Unsuccessful right-sided AVNRT ablation: Patients with unsuccessful right-sided slow pathway ablation attempt, will be candidates for Coronary sinus / left-sided slow pathway ablation.
  Interventions: Procedure: Coronary sinus / left-sided slow pathway ablation

INTERVENTIONS:
Procedure: Coronary sinus / left-sided slow pathway ablation — Patients with unsuccessful right-sided slow pathway ablation attempt will undergo a stepwise:
  1. coronary sinus slow pathway ablation, which, if unsuccessful, will be followed by
  2. left-sided slow pathway ablation, using trans-septal approach.

SUMMARY:
This proposal aims to evaluate safety and efficacy aspects of a new protocol for AVNRT ablation, using a stepwise anatomical approach.

The investigators hypothesize that the use of a standardized electro-anatomical guided strategy, using a sequential approach as follows:

1. Right-side postero-septal tricuspid annulus
2. Coronary sinus
3. Left-side postero-septal mitral annulus

For slow pathway AVNRT ablation is safe and efficient, increasing the chance of a successful ablation in difficult cases, while reducing the need of re-do procedures and the risk for high-degree atrio-ventricular block.

The investigators aim to define and implement a new standardized protocol for AVNRT ablation while at the same time assessing the efficacy and safety of coronary sinus and left-side approaches for slow-pathway ablation.

DETAILED DESCRIPTION:
Atrio-ventricular nodal reentrant tachycardia (AVNRT) is the most common form of supraventricular tachycardia in adults. The substrate of AVNRT is dual nodal atrio-ventricular (AV) physiology represented by the presence of slow (SP) and fast pathway (FP) conduction. Selective radiofrequency (RF) ablation of the slow AV nodal pathway can cure the arrhythmia with acute success rates varying from 95 to 98% and low recurrence rates during long-term follow-up.

The compact AV node sends two posterior extensions with node-like tissue distributed towards the coronary sinus and tricuspid annulus (right posterior extension) and towards the mitral annulus (left posterior extension). Earlier literature suggested that the right posterior nodal extension is involved in the tachycardia circuit of most patients with AVNRT (slow pathway input). The tachycardia circuit may rarely involve the left posterior nodal extension, in which case a left-sided ablation procedure is needed. The right-sided approach is sufficient for the majority of cases and represents today the standard protocol for AVNRT ablation.

Lee et Al., in view of current anatomical and electrophysiological knowledge concerning the AV node, proposed the following sequential approach for SP ablation:

I. the isthmus between tricuspid annulus and coronary sinus ostium (the usual site of slow pathway), II. the tricuspid edge of coronary sinus ostium (by moving the ablation catheter tip slightly in and out of the coronary sinus), III. the septum lower than coronary sinus ostium, moving higher up on the half of Koch's triangle along the septum, IV. one or two burns inside the first few centimeters of the coronary sinus, V. left side of the septum (last).

The investigators hypothesize that the use of a standardized electro-anatomical guided strategy, using a sequential approach as follows:

1. Right-side postero-septal tricuspid annulus
2. Coronary sinus
3. Left-side postero-septal mitral annulus

for slow pathway AVNRT ablation is safe and efficient, increasing the chance of a successful ablation in difficult cases, while reducing the need of re-do procedures and the risk for high-degree atrio-ventricular block.

The protocol will be applied in all patients undergoing slow pathway ablation for typical AVNRT. Those with unsuccessful right-sided attempt and who undergo coronary sinus and left-sided ablation attempt will be eligible for registry inclusion.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 and <80 years
2. History of symptomatic PSVT
3. Signed informed consent
4. Documented AVNRT during EPS with at least 1 of the following:

   * Previous unsuccessful right-sided ablation attempt
   * Ideal SP electrogram at XR < 10 mm in RAO 30°
   * Right-sided ablation attempt with:

     * VA block during JB or
     * A minimum of 7 unsuccessful RF energy deliveries, with no upper limit (to the 1st operator's discretion)

Exclusion Criteria:

* Previous CVA
* Severe mitral or aortic valve disease
* Documented intra-cardiac thrombus

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Symptomatic AVNRT patients undergoing ablation procedure
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2014-09; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Slow pathway modification/elimination | Up to 6 hours
  Success of the ablation determined at the end of the procedure, defined as slow pathway modification (persistence of AH jump with maximum of 1 echo under Isoprenaline) or elimination (No AH jump; no echo), resulting in arrhythmia non-inducibility

SECONDARY OUTCOMES:
Time to AVNRT recurrence | Up to 6 Months
  Arrhythmia (AVNRT) recurrence evaluation at routine 6-month follow-up visit, defined as: ECG/Holter documented supraventricular regular tachycardia, with/without need for re-intervention.
High-degree AV block requiring permanent pace-maker | Up to 48 hours
  Major adverse event usually occuring during ablation procedure or as late as 48 hours after the procedure
Cardiac tamponade | Up to 48 hours
  Major adverse event resulting in significant pericardial effusion with hemodynamic instability (Systolic Blood pressure <90 mmHg), requiring intervention (pericardiocentesis; cardiac surgery)
Systemic embolic events | Up to 48 hours
  Major adverse event secondary to systemic thromboembolism resulting in stroke or transient ischemic attack, or peripheral acute ischemia syndrome.
Transient AV conduction disturbance | Up to 48 hours
  Minor adverse event resulting in transient prolongation of AV conduction, transient 2nd or 3rd degree AV block.
Peripheral arterio-venous complications | Up to 48 hours
  Minor adverse event implicating the site of vascular approach, resulting in local hematoma of the groin or femoral arterio-venous fistula.
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | Up to 48 hours
  Composite endpoint for safety using previously stated adverse events: high-degree AV block requiring permanent pace-maker, cardiac tamponade, systemic embolic events, transient AV conduction disturbances, peripheral arterio-venous complications.

CONTACTS AND LOCATIONS:
Overall Officials: Roy Beinart, MD, Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McGuire MA, Robotin M, Yip AS, Bourke JP, Johnson DC, Dewsnap BI, Grant P, Uther JB, Ross DL. Electrophysiologic and histologic effects of dissection of the connections between the atrium and posterior part of the atrioventricular node. J Am Coll Cardiol. 1994 Mar 1;23(3):693-701. doi: 10.1016/0735-1097(94)90756-0. PMID 8113554
- [Background] Inoue S, Becker AE. Posterior extensions of the human compact atrioventricular node: a neglected anatomic feature of potential clinical significance. Circulation. 1998 Jan 20;97(2):188-93. doi: 10.1161/01.cir.97.2.188. PMID 9445172
- [Background] Kilic A, Amasyali B, Kose S, Aytemir K, Celik T, Kursaklioglu H, Iyisoy A, Ozmen N, Yuksel C, Lenk MK, Isik E. Atrioventricular nodal reentrant tachycardia ablated from left atrial septum: clinical and electrophysiological characteristics and long-term follow-up results as compared to conventional right-sided ablation. Int Heart J. 2005 Nov;46(6):1023-31. doi: 10.1536/ihj.46.1023. PMID 16394598
- [Background] Katritsis DG, Giazitzoglou E, Zografos T, Ellenbogen KA, Camm AJ. An approach to left septal slow pathway ablation. J Interv Card Electrophysiol. 2011 Jan;30(1):73-9. doi: 10.1007/s10840-010-9527-z. Epub 2010 Dec 14. PMID 21153692
- [Background] Lee PC, Chen SA, Hwang B. Atrioventricular node anatomy and physiology: implications for ablation of atrioventricular nodal reentrant tachycardia. Curr Opin Cardiol. 2009 Mar;24(2):105-12. doi: 10.1097/HCO.0b013e328323d83f. PMID 19225293